CLINICAL TRIAL: NCT01641562
Title: Diagnosis and Prediction of Subclinical Cardiac Dysfunction Induced by Therapy With Taxanes in Patients With Breast Cancer
Brief Title: Diagnosis and Prediction of Taxanes Induced Cardiac Dysfunction
Acronym: CARDIOTAX
Status: Completed | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Dragos Vinereanu, Professor, MD, PhD, Carol Davila University of Medicine and Pharmacy
Other Study IDs: 4192910; 112/27.10.2011 (Other Grant/Funding Number: UEFISCDI ROMANIA)
Record Dates: First submitted 2012-07-04; First posted 2012-07-17 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: BREAST CANCER,; TAXANES,; SUBCLINICAL CARDIAC DYSFUNCTION ,; DIAGNOSTIC TOOLS,; PREDICTIVE MODELS
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biomarkers: brain natriuretic peptides, troponin T, markers of myocardial fibrosis (β cross laps and procollagen type-1 amino terminal), and markers of inflammation (PCR-hs, IL1, IL6, IL 10, TNFalpha).
  Markers of the oxidative stress: concentration of carbonyl in plasmatic proteins, and the antioxidant capacity of plasma.
  Genetic tests of susceptibility to cardiotoxicity: genomic DNA extraction kit/DNA quantification tests/PCR tests.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TAXANES: patients with early breast cancer, scheduled to receive taxanes, with doses according to the stage of the disease

SUMMARY:
Breast cancer represents the most frequent form of neoplasia in women worldwide, being responsible of 1.6% of annual deaths. Therefore, it is a major public health issue and research in this field should be a priority. Taxanes, such as paclitaxel and docetaxel, are extremely powerful antineoplastic drugs, which alone or in association to anthracyclines, increase survival and lower the recurrence rate of cancer, but their use is limited by cardiotoxicity. Cardiotoxicity can appear early or late after therapy, and may vary from subclinical myocardial dysfunction to irreversible heart failure. Currently, cardiac dysfunction induced by taxanes is diagnosed through classical echocardiographic parameters. However, these cannot detect subtle, early changes of cardiac structure and function. Consequently, description of new parameters, which could detect cardiac dysfunction in an early stage, becomes essential for detecting the group of patients at risk for irreversible heart failure. The objectives of the investigators project, in patients with breast cancer treated with taxanes, are to investigate their mechanisms which lead to cardiac dysfunction, to describe new parameters for the early diagnosis of cardiotoxicity, and to define predictive models for cardiotoxicity. Meanwhile, project will publish the results in prestigious journals, leading to an increase of the visibility of Romanian research internationally.

DETAILED DESCRIPTION:
Scientific context and motivation. Breast cancer represents the most frequent form of neoplasia in women worldwide, comprising 16% off all neoplasias. A report of the World Health Organization showed that 1 from 6 cancers is determined by breast cancer and this form of neoplasm causes around 550,000 deaths/year, respective 1.6% of all annual deaths in the world. The incidence of breast cancer is increasing, over 1.1 million of women being newly diagnosed with cancer every year. Although considered a pathology specific to developed countries, recently it was established that developing countries, such as Romania, include over 69% of all breast cancers. Therefore, breast cancer is currently a major public health and economical issue and research on new therapies, as well as monitoring their safety use, should be a priority.

Many studies showed that, due to new chemotherapy, breast cancer can be considered a curable disease. And indeed, use of a multidisciplinary approach - surgery, radiotherapy, chemotherapy - has conducted to a significant reduction in the mortality. As a consequence of increased life expectancy, it becomes essential that specific oncologic therapies should be safe.

Taxanes, inhibitors of cellular mitosis (paclitaxel and docetaxel), relatively new drugs, are extremely potent and widely used in different therapeutic regimes. Their single use or the association with classical chemotherapy, have been proved to increase significantly rate of cure in breast cancer, as well as to reduce recurrences. However, the applicability of these drugs on medium or long term is limited by the risk of cardiotoxicity.

Cardiotoxicity is one of the most important adverse reactions of taxanes, leading to an important increase of morbidity and mortality. Cardiotoxicity can appear early or late in the course of the disease, and may vary from subclinical myocardial dysfunction to irreversible heart failure or even death. Recent research has showed that cardiac dysfunction induced by taxanes may increase exponentially with the cumulative dose used; meanwhile, it may be augmented by other associated cytotoxic drugs. Data on the susceptibility of patients to develop cardiotoxicity are scarce. Some studies suggest that patients without known cardiovascular history may develop symptomatic heart failure in direct connection to the cumulative dose received, affirmation which has led to the use of reduced doses of chemotherapy and, therefore, to a reduction in their efficiency. But also under these circumstances, there is a risk of cardiotoxicity induced by taxanes therapy, risk which cannot be foreseen by the cumulative dose. Moreover, the cardiac alteration is very frequently subclinical and it can appear early (during therapy), late (during the first year after therapy) or very late (more than one year after finishing therapy). Consequently, early diagnosis of subclinical cardiac dysfunction in patients with breast cancer treated with taxanes, as well as the establishment of prediction models for irreversible heart failure is essential in the management of such patients.

Currently, recommendations of diagnosis of cardiac dysfunction induced by taxanes are to use functional and structural parameters of conventional echocardiography, such as left ventricular ejection fraction (LVEF), left ventricular shortening fraction (LVSF), as well as diameters and volumes of the heart chambers. However, sometime, these conventional measurements allow only the late diagnosis of cardiac dysfunction, which might be already irreversible. Therefore, description of new and simple parameters, able to diagnose more subtle, subclinical changes of cardiac function becomes mandatory.

Recently, it has been showed that myocardial velocities, cardiac deformation, parameters of ventricular torsion, and parameters of intra- and inter- ventricular dyssynchrony are affected before reduction of LVEF and LVSF. Therefore, these parameters might be useful in the early diagnosis of cardiac dysfunction induced by taxanes, and in establishing prediction of cardiotoxicity.

Meanwhile, recently, early diagnosis of cardiac dysfunction is also based on increase of the biomarkers. Some of them, such as such as brain natriuretic peptides, troponins, markers of cardiac fibrosis and inflammation, might be more important during the subclinical cardiac dysfunction induced by chemotherapy, hypothesis that will be also verified.

Finally, it was suggested that therapy with taxanes might increase the oxidative stress, causing endothelial dysfunction with increased arterial stiffness. This might be a mechanisms by which taxanes promotes cardiac dysfunction, through alteration of ventriculo-arterial coupling.

In conclusion, early detection of cardiovascular dysfunction and establish of predictive models for cardiotoxicity represent a priority in the management of breast cancer. This can be done by using new ultrasound technique, assessing subclinical myocardial disease and ventriculo-arterial coupling, and new laboratory methods, assessing different biomarkers and the oxidative stress.

Objectives. The main objective of our project is to describe new parameters for the early diagnosis of cardiovascular dysfunction patients with early breast cancer, treated with taxanes, and to define predictive models for cardiotoxicity.

Our hypotheses are based on:

1. Taxanes (alone or in combination with anthracycline) increase oxidative stress, with excessive production of free oxygen radicals, and activation of neurohormonal mediators of inflammation and fibrosis. Decrease of antioxidant capacity, genetically determined, might be an additional mechanism is some patients. Therefore, we will test the hypothesis that imbalance between oxidative stress and antioxidant capacity is one of the main mechanism of cardiotoxicity induced by taxanes in patients with breast cancer.
2. Oxidative stress determines endothelial dysfunction with arterial remodeling and increased arterial stiffness. We will test the hypothesis that impaired endothelial-arterial-ventricular coupling might play an important role in the cardiotoxicity induced by chemotherapy.
3. Subclinical cardiac dysfunction can be diagnosed by looking to new parameters of myocardial deformation and torsion, and their timing into the cardiac cycle. We assume that these parameters are first affected, before conventional echo parameters, during cardiotoxicity induced by chemotherapy.

Therefore, objectives of our study, in patients with early breast cancer, without cardiovascular symptoms, treated with taxanes (alone or in combination with anthracycline), are:

1. To assess imbalance between oxidative stress and antioxidant capacity in order to describe new potential mechanisms of cardiotoxicity;
2. To test implication of some genetic disorders in predicting cardiotoxicity, mainly through decrease of antioxidant capacity;
3. To assess endothelial-arterial-ventricular coupling as a possible determinant of cardiotoxicity;
4. To determine the diagnostic accuracy of new echo parameters, as well as new biomarkers, for the early diagnosis of cardiotoxicity.
5. To establish a standard evaluation protocol, by using these parameters and their predictive value, in order to identify patients at risk.

By achieving these objectives of our research, derived objectives are:

1. To promote original research in a new and important interdisciplinary field (cardiotoxicity induced by chemotherapy);
2. To increase international visibility of Romanian research by publishing the results;
3. To increase the research capacity of our unit, also by attracting new researchers;
4. To further develop an interdisciplinary research center, attached to our new oncology unit; to participate to international muticentric studies/networks in the cardio-oncology field.

Method and approach. Study population. Study will include 60 patients with early breast cancer, scheduled to receive taxanes, in monotherapy (30 patients) or associated to anthracyclines (30 patients), with doses according to the stage of the disease. Inclusion criteria are: (1) Age over 18 years; (2) Informed consent signed; (3) Patients with early breast cancer, scheduled to receive chemotherapy; (4) LVEF > 50% and LVSF > 20%. Exclusion criteria are: (1) Any history of cardiovascular disease and/or active cardiovascular treatment; (2) Diabetes mellitus; (3) Mediastinal irradiation. The protocol will be sent for approval to the Local Ethic Committee. All patients referred to the oncology department with the diagnosis of breast cancer, and scheduled to receive chemotherapy, will be screened. Patients will be evaluated 24 hours before initiation of treatment, and within 24 hours from the end of the cycle of chemotherapy. Long-term follow-up will be performed at 1 and 2 years after the end of chemotherapy.

Methods. All patients will be assessed by:

1. General characteristics: age, sex, height, weight, blood pressure, heart rate, family history, risk factors, clinical stage of breast cancer, date of surgical intervention (if applicable), date of initiation of chemotherapy, details of the scheme of chemotherapy, etc.
2. Electrocardiogram (12 leads) and routine blood samples.
3. Biomarkers: brain natriuretic peptides, troponin T, markers of myocardial fibrosis (β cross laps and procollagen type-1 amino terminal), and markers of inflammation (PCR-hs, IL1, IL6, IL 10, TNFalpha).
4. Markers of the oxidative stress: concentration of carbonyl in plasmatic proteins, and the antioxidant capacity of plasma.
5. Genetic tests of susceptibility to cardiotoxicity: genomic DNA extraction kit/DNA quantification tests/PCR tests.
6. Echocardiography: detailed echo examination (VIVID 7 GE echo machine, with dedicated software ECHOPAC BT09) will be performed, as follows:

   1. Conventional echocardiography will measure/calculate:

      * Structural parameters: thickness of the cardiac walls; diameters and volumes of the cardiac cavities, aorta, and pulmonary artery; left ventricular mass; relative wall thickness; wall stress.
      * Functional parameters of systolic and diastolic function: ejection fraction, shortening fraction, stroke volume, cardiac output, cardiac index, tricuspid and mitral annular excursions; and, respectively, parameters derived from the transmitral flow, pulmonary veins flow, velocity of propagation of the mitral flow into the LV.
   2. Q analysis by tissue velocity imaging: measurements of systolic and diastolic myocardial velocities, and of the isovolumic accelerations, at the level of multiple left and right ventricular myocardial segments.
   3. Speckle tracking imaging, which is a new non-invasive method for the assessment of cardiac global and regional function; it uses myocardial speckles that represent tissue markers that can be tracked frame by frame throughout the cardiac cycles. Motion is analyzed by integrating frame by frame changes. This new method offers an alternative to techniques such as color-coded tissue velocity imaging for myocardial deformation (measured as strain and strain rate) in radial, longitudinal, and circumferential directions, in order to assess left and right ventricular, systolic and diastolic function, left ventricular torsion, and left and right atrial function.
   4. Advanced Q-Scan imaging, which is a new and innovative dedicated parametric imaging, supported by the 4D probe, for quantitative display of regional wall deformation. It consists of tissue synchronization, a real time parametric imaging technique for displaying mechanical synchronicity, and strain and strain rate imaging, showing myocardial deformation and the rate of deformation in real time.
   5. 3D echocardiography allows precise evaluation of the cardiac chamber anatomy and function. 4D analysis enables post-processing of multi-plane imaging datasets, allows multi-dimensional imaging acquired in parasternal bi-plane and apical tri-plane views, and supports 2D, color, as well as, tissue Doppler modes (including tissue synchronization imaging). All data can be stored in raw data DICOM format and can be recalled for post-processing.
7. Measurement of endothelial function, parameters of arterial remodeling, and arterial stiffness at the level of the common carotid artery (vascular remodeling and arterial stiffness indices), and at the level of the brachial artery (endothelial function). Assessment will be done using an ALOKA α10 ultrasound machine, using a high resolution probe of 7,5-10 MHz, equipped with an "echo-tracking" system. Meanwhile, a dedicated new software available on the machine (wave intensity analysis) will be used to assess ventriculo-arterial coupling. Another system (Complior) will be used in order to measure the pulse wave velocity between 2 arterial sites (carotid-femoral and carotido-radial), as another measure of arterial stiffness.

The research team who will participate in the project has an important experience in the field of cardiology and use of the new ultrasound techniques, as well as in the field of oncology, especially breast cancer, with many publications, national and international communications/ lectures on these topics.

The Working Plan is well adapted for achieving the goals of this project, and human and material resources are appropriate to achieve all the objectives of the projects, taking into account the existing and newly acquired resources and infrastructure.

Impact, relevance, applications. The relevance for the field. Because breast cancer is the most frequent neoplasia in women worldwide, including Romania, and the most feared adverse effect of chemotherapy is cardiac dysfunction, which leads to a significant increase in morbidity, mortality, and economical costs, we believe that the identification in early stages of cardiac dysfunction is a health problem of major interest and should represent a priority of the cardiology and oncology research. Using new imagistic and laboratory parameters might allow their integration into predictive scores, essential to identify patients at risk and to optimize treatment strategies in these patients.

The estimated impact and applications of the project. This project could contribute to the elucidation of mechanisms of cardiac dysfunction induced by taxanes (alone or in combination with anthracyclines). Moreover, it might be able to introduce into clinical practice new diagnostic and predictive methods for patients at risk for developing cardiac dysfunction, consequently leading to an optimization of chemotherapy. Therefore, the results of the project could be applicative also from social and economic purposes, taking into account the disabilities and costs of heart failure that could occur after chemotherapy. Our proposal fits into the strategic objectives of our National System of Exploratory Research Projects, initiated by CNCSIS. It will create knowledge in the medical field and generate important scientific results, nationally and internationally competitive.

The results of the project might be able to generate:

1. Publication of results in prestigious, ISI indexed journals, contributing to the rise of the visibility of Romanian research at international level;
2. Increase of the research capacity of our unit, also by attracting new researchers, which will have the chance to complete their training in an adequate scientific environment;
3. A national interdisciplinary (cardiology and oncology) network dedicated to the early diagnostic and prediction of cardiotoxicity;
4. The premises of interdisciplinary, national and international collaboration, with other centers with common interest, collaboration which could be the background of new research projects.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Informed consent signed
3. Patients with early breast cancer, scheduled to receive chemotherapy
4. LVEF > 50% and LVSF > 20%.

Exclusion Criteria:

1. Any history of cardiovascular disease and/or active cardiovascular treatment
2. Diabetes mellitus
3. Mediastinal irradiation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will include 60 patients with early breast cancer, scheduled to receive taxanes, in monotherapy (30 patients) or associated to anthracyclines (30 patients), with doses according to the stage of the disease.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-01-01; Primary Completion 2016-10-30 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
CARDIOTOXICITY PREDICTION SCORE | 6 MONTHS, 1 YEAR, 2 YEARS
  To determine the change in left ventricular ejection fraction (LVEF) after 6 months, 1 or 2 years after treatment with taxanes for defining cardiotoxicity (LVEF less than 55% or reduction with more than 10% from baseline).

SECONDARY OUTCOMES:
GENETIC DISORDERS AND CARDIOTOXICITY | BASELINE
  To test implication of some genetic disorders in predicting cardiotoxicity, mainly through decrease of antioxidant capacity;
DIAGNOSTIC ACCURACY FOR CARDIOTOXICITY | 2 YEARS
  Diagnostic accuracy of new echo parameters, as well as new biomarkers, for the early diagnosis of cardiotoxicity.
EVALUATION PROTOCOL FOR CARDIOTOXICITY | 2 YEARS
  To establish a standard evaluation protocol, by using these parameters and their predictive value, in order to identify patients at risk for cardiac dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: DRAGOS VINEREANU, MD, Study Director — UNIVERSITY AND MEDICINE CAROL DAVILA BUCHAREST
Locations (1):
- University and Emergency Hospital, Bucharest, Romania